CLINICAL TRIAL: NCT01496885
Title: A Multicenter Observational Study to Evaluate the Simplified STroke REhabilitation Assessment of Movement (S-STREAM) Scale in Subjects Obtained Between 24 and 48 Hours of a Nonhemorrhagic Ischemic Stroke
Brief Title: Observational Study to Evaluate the Simplified-STroke REhabilitation Assessment of Movement (S-STREAM) Scale in Subjects Who Have Experienced a Nonhemorrhagic Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: ASBI 801
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Nonhemorrhagic Ischemic Stroke; Motor Function
Keywords: stroke
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nonhemorrhagic Ischemic Stroke: Subjects obtained within 24 to 48 hours of a nonhemorrhagic ischemic stroke
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This was an observational study and no study drug was administered.

SUMMARY:
The purpose of this study is to evaluate the utility of the S-STREAM as an instrument to assess motor function in subjects who have experienced a nonhemorrhagic ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 21 and 85 years, inclusive
* Participants had no prior history of stroke (unless the stroke was silent or not associated with a motor deficit) presented between 24 and 48 hours from onset with an acute stroke with clinical assessments and imaging studies (conducted as part of the standard of care procedures in stroke patients) indicating that the stroke was ischemic, with no secondary hemorrhage large enough to exert a mass effect that would contribute significantly to the neurological deficit (small punctate hemorrhages were permitted), in the vascular distribution of the middle cerebral artery and not classifiable as a lacunar stroke
* Participants understood and agreed to comply with the requirements of the study and they were willing to provide verbal/nonverbal informed consent indicating voluntary consent to participate in the study
* Participants were to have scored at least 16 on the Mini Mental Status Examination (MMSE) at screening. If the participant had an expressive aphasia and was unable to qualify based on the MMSE, the participant may have been evaluated with a language-modified form of the MMSE1 in conjunction with the investigator's clinical assessment that the participant was cognitively able to complete study procedures and stroke scales to determine eligibility. If the aphasia was too severe for the participant to complete the language-modified MMSE, the participant was excluded.
* Participants had to have a total score between 20 and 85, inclusive, on the S-STREAM administered between 24 and 48 hours after stroke onset

Exclusion Criteria:

* History of previous stroke; uncontrolled severe hypertension; dementia; advanced Parkinson disease or other significant movement disorders; or other clinically significant diseases which, in the opinion of the investigator, would have jeopardized the safety of the participant or impacted the validity of the study results
* Development of hemodynamic instability following the stroke as manifested by a persistent post stroke systolic blood pressure less than 80 mm Hg (or was dependent on medications to maintain a systolic blood pressure greater than or equal to 80 mm Hg) or greater than 190 mm Hg at the time of screening
* Presence of significant global or receptive aphasia that would have interfered with the participant's ability to understand and comply with study procedures or complete stroke assessments
* Abnormal clinical laboratory values on routine clinical laboratory test values at screening including alanine transaminase or aspartate transaminase greater than or equal to 3 times the upper limit of normal, serum creatinine greater than or equal to 3.0 mg/dL, or hemoglobin less than or equal to 10 g/dL, or any other laboratory investigation deemed by the investigator to be indicative of a clinically significant illness that could have prevented the participant from complying with study procedures or impacted on the outcome of the stroke scales
* History of drug or alcohol abuse
* History of any surgery or presence of any medical condition that, in the judgment of the investigator, may have affected the validity of the study results
* Current participation in another clinical study involving administration of an investigational product or history of such participation within 30 days of screening
* Unable to complete baseline S-STREAM and NIHSS assessments within 48 hours of stroke onset

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants may be selected upon admission to an acute care emergency center, inpatient facility, or rehabilitation center.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-01-18 (Actual); Primary Completion 2013-05-22 (Actual); Study Completion 2013-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (25):
- United States (21):
  - Newport Beach, California
  - Englewood, Colorado
  - Lawrenceville, Georgia
  - Chicago, Illinois
  - Des Moines, Iowa
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Edison, New Jersey
  - Brooklyn, New York
  - The Bronx, New York
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Canada (4):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Greenfield Park, Quebec
  - Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 120 participants who met all inclusion and no exclusion criteria were enrolled in the study at 36 sites (30 sites in the United States and 6 sites in Canada).
Pre-assignment Details: All participants received standard of care based on investigator opinion and institutional policy.
Groups:
- All Participants: Participants who were obtained within 24 to 48 hours of a nonhemorrhagic ischemic stroke.
Period: Overall Study
Arm/Group | All Participants
Started | 120
Completed | 97
Not Completed | 23
Not completed — Lost to Follow-up | 13
Not completed — Withdrawal by Subject | 7
Not completed — Clinically significant change in subject status that prevented compliance or impacted stroke outcome | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Primary Analysis population.
Arm/Group | All Participants
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (13.3)
Age, Customized [Median (Full Range); unit: years] | 67.0 [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 103
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 35
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Simplified-STroke Rehabilitation Assessment of Movement (S-STREAM) Score in Participants Obtained Between 24 and 48 Hours of a Non-hemorrhagic Ischemic Stroke
Description: The S-STREAM is composed of 5 items each across 3 components (upper limb movements, lower limb movements, and mobility). Limb movements are scored on a scale ranging from 0 (unable to perform) to 2 (able to complete the movement comparable to the unaffected side). Basic mobility items are scored on a scale ranging from 0 (unable to perform) to 3 (able to complete the activity). All S-STREAM scores were transformed to a range of 0 to 100 via Rasch transformation since the S-STREAM fit the requirements of the Rasch model. The raw scores were Rasch transformed to achieve logits scores and then remapped from the logit score to a 0 to 100 scale, where 0 indicates worst outcome and 100 indicate best outcome.
  The mean change from baseline in S-STREAM Rasch-transformed score is being reported; higher S-STREAM scores indicate better outcomes.
Time Frame: Baseline up to Day 84 post non-hemorrhagic ischemic stroke
Population: Total Simplified-Stroke Rehabilitation Assessment of Movement (S-STREAM) score was assessed in the Primary Analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 120
score on a scale
  Baseline | 57.6 (15.97)
  Day 3: number analyzed (Participants) | 113
  Day 3 | 60.9 (19.77)
  Day 7: number analyzed (Participants) | 113
  Day 7 | 66.3 (22.79)
  Day 28: number analyzed (Participants) | 101
  Day 28 | 77.4 (22.57)
  Day 56: number analyzed (Participants) | 95
  Day 56 | 80.0 (20.82)
  Day 84: number analyzed (Participants) | 97
  Day 84 | 83.0 (19.35)
  Change from baseline to Day 3: number analyzed (Participants) | 113
  Change from baseline to Day 3 | 4.2 (9.59)
  Change from baseline to Day 7: number analyzed (Participants) | 113
  Change from baseline to Day 7 | 8.9 (13.39)
  Change from baseline to Day 28: number analyzed (Participants) | 101
  Change from baseline to Day 28 | 19.5 (16.50)
  Change from baseline to Day 56: number analyzed (Participants) | 95
  Change from baseline to Day 56 | 22.7 (17.05)
  Change from baseline to Day 84: number analyzed (Participants) | 97
  Change from baseline to Day 84 | 24.8 (16.39)

2. Primary Outcome: Mean Percent Change From Baseline in Total Simplified-STroke Rehabilitation Assessment of Movement (S-STREAM) Score in Participants Obtained Between 24 and 48 Hours of a Non-hemorrhagic Ischemic Stroke
Description: The S-STREAM is composed of 5 items each across 3 components (upper limb movements, lower limb movements, and mobility). Limb movements are scored on a 3-point integer scale ranging from 0 (unable to perform) to 2 (able to complete the movement comparable to the unaffected side). Basic mobility items are scored on a 4-point integer scale ranging from 0 (unable to perform) to 3 (able to complete the activity). All S-STREAM scores were transformed to a range of 0 to 100 via Rasch transformation since the S-STREAM has been shown to fit the requirements of the Rasch model. The raw scores were Rasch transformed to get the logits scores and then remapped from the logit score to a 0 to 100 scale, where 0 indicates worst outcome and 100 indicate best outcome.
  The mean percent change from baseline in S-STREAM Rasch transformed score is being reported; higher S-STREAM scores indicate better outcomes.
Time Frame: Baseline up to Day 84 post non-hemorrhagic ischemic stroke
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | All Participants
Number analyzed (Participants) | 113
percent change
  Day 3 | 6.9 (20.18)
  Day 7 | 15.0 (26.92)
  Day 28: number analyzed (Participants) | 101
  Day 28 | 37.3 (40.78)
  Day 56: number analyzed (Participants) | 95
  Day 56 | 45.6 (43.40)
  Day 84: number analyzed (Participants) | 97
  Day 84 | 49.7 (47.00)

3. Primary Outcome: Number of Participants Obtained Between 24 and 48 Hours of a Non-hemorrhagic Ischemic Stroke With Total Simplified-STroke Rehabilitation Assessment of Movement (S-STREAM) Score, by Category
Description: The S-STREAM is composed of 5 items each across 3 components (upper limb movements, lower limb movements, and mobility). The S-STREAM assessments are conducted in the order of the following positions: supine, sitting, and standing. Limb movements are scored on a 3-point integer scale ranging from 0 (unable to perform) to 2 (able to complete the movement comparable to the unaffected side). Basic mobility items are scored on a 4-point integer scale ranging from 0 (unable to perform) to 3 (able to complete the activity). Based on the point scales described, the maximum score for upper limb movements is 10, for lower limb movements is 10, and for mobility is 15; the maximum aggregate S-STREAM raw score is therefore 35. Higher S-STREAM scores indicated better outcome. Total S-STREAM scores were generated using Rasch transformations and subsequently scaled to scores between 0 and 100 for purposes of analysis with higher total S-STREAM scores indicating a better outcome.
Time Frame: Baseline up to Day 84 post non-hemorrhagic ischemic stroke
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 120
Participants
  Baseline: 0 to <20 score | 1
  Baseline: 20 to <50 score | 38
  Baseline: 50 to <70 score | 51
  Baseline: ≥70 score | 30
  Day 3: 0 to <20 score: number analyzed (Participants) | 113
  Day 3: 0 to <20 score | 3
  Day 3: 20 to <50 score: number analyzed (Participants) | 113
  Day 3: 20 to <50 score | 22
  Day 3: 50 to <70 score: number analyzed (Participants) | 113
  Day 3: 50 to <70 score | 45
  Day 3: ≥70 score: number analyzed (Participants) | 113
  Day 3: ≥70 score | 43
  Day 7: 0 to <20 score: number analyzed (Participants) | 113
  Day 7: 0 to <20 score | 3
  Day 7: 20 to <50 score: number analyzed (Participants) | 113
  Day 7: 20 to <50 score | 19
  Day 7: 50 to <70 score: number analyzed (Participants) | 113
  Day 7: 50 to <70 score | 35
  Day 7: ≥70 score: number analyzed (Participants) | 113
  Day 7: ≥70 score | 56
  Day 28: 0 to <20 score: number analyzed (Participants) | 101
  Day 28: 0 to <20 score | 5
  Day 28: 20 to <50 score: number analyzed (Participants) | 101
  Day 28: 20 to <50 score | 6
  Day 28: 50 to <70 score: number analyzed (Participants) | 101
  Day 28: 50 to <70 score | 17
  Day 28: ≥70 score: number analyzed (Participants) | 101
  Day 28: ≥70 score | 73
  Day 56: 0 to <20 score: number analyzed (Participants) | 95
  Day 56: 0 to <20 score | 1
  Day 56: 20 to <50 score: number analyzed (Participants) | 95
  Day 56: 20 to <50 score | 9
  Day 56: 50 to <70 score: number analyzed (Participants) | 95
  Day 56: 50 to <70 score | 12
  Day 56: ≥70 score: number analyzed (Participants) | 95
  Day 56: ≥70 score | 73
  Day 84: 0 to <20 score: number analyzed (Participants) | 97
  Day 84: 0 to <20 score | 2
  Day 84: 20 to <50 score: number analyzed (Participants) | 97
  Day 84: 20 to <50 score | 6
  Day 84: 50 to <70 score: number analyzed (Participants) | 97
  Day 84: 50 to <70 score | 9
  Day 84: ≥70 score: number analyzed (Participants) | 97
  Day 84: ≥70 score | 80

4. Secondary Outcome: Subgroup Analysis of Total S-STREAM Score and Mean Change From Baseline to Day 84 in Participants Obtained Between 24 and 48 Hours of a Non-hemorrhagic Ischemic Stroke
Description: The S-STREAM is composed of 5 items each across 3 components (upper limb movements, lower limb movements, and mobility). Limb movements are scored on a 3-point integer scale ranging from 0 (unable to perform) to 2 (able to complete the movement comparable to the unaffected side). Basic mobility items are scored on a 4-point integer scale ranging from 0 (unable to perform) to 3 (able to complete the activity). All S-STREAM scores were transformed to a range of 0 to 100 via Rasch transformation since the S-STREAM has been shown to fit the requirements of the Rasch model. The raw scores were Rasch transformed to get the logits scores and then remapped from the logit score to a 0 to 100 scale, where 0 indicates worst outcome and 100 indicate best outcome.
  The mean change from baseline in S-STREAM Rasch-transformed score is being reported; higher S-STREAM scores indicate better outcomes.
Time Frame: Baseline up to Day 84 post non-hemorrhagic ischemic stroke
Population: Subgroup analysis of Total Simplified-STroke Rehabilitation Assessment of Movement (S-STREAM) score was assessed in patients with available data in the Primary Analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 104
score on a scale
  Baseline: USA: number analyzed (Participants) | 85
  Baseline: USA | 58.7 (14.80)
  Baseline: Canada: number analyzed (Participants) | 35
  Baseline: Canada | 55.0 (18.49)
  Day 84: USA: number analyzed (Participants) | 66
  Day 84: USA | 82.7 (18.35)
  Day 84: Canada: number analyzed (Participants) | 31
  Day 84: Canada | 83.7 (21.63)
  Change from baseline: United States: number analyzed (Participants) | 66
  Change from baseline: United States | 23.1 (16.04)
  Change from baseline: Canada: number analyzed (Participants) | 31
  Change from baseline: Canada | 28.4 (16.82)
  Baseline: <75 years: number analyzed (Participants) | 89
  Baseline: <75 years | 58.1 (16.56)
  Baseline: ≥75 years: number analyzed (Participants) | 31
  Baseline: ≥75 years | 56.2 (14.27)
  Day 84: <75 years: number analyzed (Participants) | 72
  Day 84: <75 years | 84.9 (19.74)
  Day 84: ≥75 years: number analyzed (Participants) | 25
  Day 84: ≥75 years | 77.6 (17.44)
  Change from baseline: <75 years: number analyzed (Participants) | 72
  Change from baseline: <75 years | 26.4 (17.33)
  Change from baseline: ≥75 years: number analyzed (Participants) | 25
  Change from baseline: ≥75 years | 20.2 (12.54)
  Baseline: Male: number analyzed (Participants) | 69
  Baseline: Male | 57.0 (15.93)
  Baseline: Female: number analyzed (Participants) | 51
  Baseline: Female | 58.5 (16.15)
  Day 84: Male: number analyzed (Participants) | 58
  Day 84: Male | 82.4 (19.70)
  Day 84: Female: number analyzed (Participants) | 39
  Day 84: Female | 83.9 (19.04)
  Change from baseline: Male: number analyzed (Participants) | 58
  Change from baseline: Male | 25.4 (16.22)
  Change from baseline: Female: number analyzed (Participants) | 39
  Change from baseline: Female | 23.9 (16.82)
  Baseline: Body mass index, <30 kg/mg^2: number analyzed (Participants) | 83
  Baseline: Body mass index, <30 kg/mg^2 | 56.3 (15.55)
  Baseline: Body mass index, ≥30 kg/mg^2: number analyzed (Participants) | 37
  Baseline: Body mass index, ≥30 kg/mg^2 | 60.6 (16.71)
  Day 84: Body mass index, <30 kg/mg^2: number analyzed (Participants) | 66
  Day 84: Body mass index, <30 kg/mg^2 | 82.9 (17.88)
  Day 84: Body mass index, ≥30 kg/mg^2: number analyzed (Participants) | 31
  Day 84: Body mass index, ≥30 kg/mg^2 | 83.2 (22.48)
  Change from baseline: Body mass index, <30 kg/mg^2: number analyzed (Participants) | 66
  Change from baseline: Body mass index, <30 kg/mg^2 | 26.5 (15.98)
  Change from baseline: Body mass index, ≥30 kg/mg^2: number analyzed (Participants) | 31
  Change from baseline: Body mass index, ≥30 kg/mg^2 | 21.2 (16.95)
  Baseline: Right handedness | 57.6 (16.01)
  Baseline: Left handedness: number analyzed (Participants) | 16
  Baseline: Left handedness | 57.9 (16.20)
  Day 84: Right handedness: number analyzed (Participants) | 85
  Day 84: Right handedness | 82.3 (18.57)
  Day 84: Left Handedness: number analyzed (Participants) | 12
  Day 84: Left Handedness | 88.2 (24.51)
  Change from baseline: Right handedness: number analyzed (Participants) | 85
  Change from baseline: Right handedness | 24.0 (16.25)
  Change from baseline: Left handedness: number analyzed (Participants) | 12
  Change from baseline: Left handedness | 30.4 (17.07)
  Baseline: Left and right side of brain affected: number analyzed (Participants) | 1
  Baseline: Left and right side of brain affected | 50.1
  Baseline: Left side of brain affected: number analyzed (Participants) | 36
  Baseline: Left side of brain affected | 59.4 (15.47)
  Baseline: Right side of brain affected: number analyzed (Participants) | 53
  Baseline: Right side of brain affected | 54.8 (17.19)
  Baseline: Unknown area of brain affected: number analyzed (Participants) | 30
  Baseline: Unknown area of brain affected | 60.6 (14.10)
  Day 84: Left and right side of brain affected: number analyzed (Participants) | 1
  Day 84: Left and right side of brain affected | 79.3
  Day 84: Left side of brain affected: number analyzed (Participants) | 29
  Day 84: Left side of brain affected | 84.2 (19.65)
  Day 84: Right side of brain affected: number analyzed (Participants) | 43
  Day 84: Right side of brain affected | 82.2 (22.98)
  Day 84: Unknown area of brain affected: number analyzed (Participants) | 24
  Day 84: Unknown area of brain affected | 83.2 (11.18)
  Change from baseline: Left and right side of brain affected: number analyzed (Participants) | 1
  Change from baseline: Left and right side of brain affected | 29.2
  Change from baseline: Left side of brain affected: number analyzed (Participants) | 29
  Change from baseline: Left side of brain affected | 24.6 (17.17)
  Change from baseline: Right side of brain affected: number analyzed (Participants) | 43
  Change from baseline: Right side of brain affected | 26.7 (17.04)
  Change from baseline: Unknown area of brain affected: number analyzed (Participants) | 24
  Change from baseline: Unknown area of brain affected | 21.4 (14.58)
  Baseline: tPA use at baseline, yes: number analyzed (Participants) | 20
  Baseline: tPA use at baseline, yes | 51.8 (15.69)
  Baseline: tPA use at baseline, no: number analyzed (Participants) | 100
  Baseline: tPA use at baseline, no | 58.7 (15.85)
  Day 84: tPA use at baseline, yes: number analyzed (Participants) | 16
  Day 84: tPA use at baseline, yes | 85.8 (18.36)
  Day 84: tPA use at baseline, no: number analyzed (Participants) | 81
  Day 84: tPA use at baseline, no | 82.5 (19.60)
  Change from baseline: tPA use at baseline, yes: number analyzed (Participants) | 16
  Change from baseline: tPA use at baseline, yes | 32.0 (14.16)
  Change from baseline: tPA use at baseline, no: number analyzed (Participants) | 81
  Change from baseline: tPA use at baseline, no | 23.4 (16.51)

5. Secondary Outcome: Mean Change From Baseline in National Institutes of Health Stroke Scale (NIHSS) Score in Participants Obtained Between 24 and 48 Hours of a Non-hemorrhagic Ischemic Stroke
Description: The NIHSS is a stroke deficit assessment scale composed of 11 components, where a score of 0 is defined as normal while higher scores indicate increasing severity of impairment for each component. Components include level of consciousness (3 evaluations, 2 of which are scored 0 to 2 and 1 of which is scored 0 to 3), best gaze (scored 0 to 2), visual (scored 0 to 3), facial palsy (scored 0 to 3), motor arm (scored 0 to 4 in both arms), motor leg (scored 0 to 4 in both legs), limb ataxia (scored 0 to 2), sensory (scored 0 to 2), best language (scored 0 to 3), dysarthria (scored 0 to 2), and extinction and inattention (scored 0 to 2). The total NIHSS score is calculated by summing individual scores. The maximum total score on the NIHSS is 42 and the level of stroke severity ranges from 0 (normal, no stroke) to 42 (severe stroke). Higher NIHSS scores indicate worse outcome.
  The mean change from baseline is also being reported; the greater the negative value, the better the outcome.
Time Frame: Baseline up to Day 84 post non-hemorrhagic ischemic stroke
Population: National Institutes of Health Stroke Scale (NIHSS) Score was assessed in the Primary Analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 118
score on a scale
  Baseline | 6.2 (3.64)
  Day 3: number analyzed (Participants) | 113
  Day 3 | 5.4 (3.81)
  Day 7: number analyzed (Participants) | 113
  Day 7 | 4.6 (3.88)
  Day 28: number analyzed (Participants) | 10
  Day 28 | 3.1 (3.57)
  Day 56: number analyzed (Participants) | 96
  Day 56 | 2.5 (2.97)
  Day 84: number analyzed (Participants) | 97
  Day 84 | 2.1 (2.85)
  Change from baseline: Day 3: number analyzed (Participants) | 113
  Change from baseline: Day 3 | -0.9 (1.77)
  Change from baseline: Day 7: number analyzed (Participants) | 113
  Change from baseline: Day 7 | -1.6 (2.49)
  Change from baseline: Day 28: number analyzed (Participants) | 10
  Change from baseline: Day 28 | -3.1 (3.56)
  Change from baseline: Day 56: number analyzed (Participants) | 96
  Change from baseline: Day 56 | -3.8 (3.42)
  Change from baseline: Day 84: number analyzed (Participants) | 97
  Change from baseline: Day 84 | -4.3 (3.09)

6. Secondary Outcome: Mean Percent Change From Baseline in National Institutes of Health Stroke Scale Score in Participants Obtained Between 24 and 48 Hours of a Non-hemorrhagic Ischemic Stroke
Description: The NIHSS is a stroke deficit assessment scale composed of 11 components, where a score of 0 is defined as normal while higher scores indicate increasing severity of impairment for each component. Components include level of consciousness (3 evaluations, 2 of which are scored 0 to 2 and 1 of which is scored 0 to 3), best gaze (scored 0 to 2), visual (scored 0 to 3), facial palsy (scored 0 to 3), motor arm (scored 0 to 4 in both arms), motor leg (scored 0 to 4 in both legs), limb ataxia (scored 0 to 2), sensory (scored 0 to 2), best language (scored 0 to 3), dysarthria (scored 0 to 2), and extinction and inattention (scored 0 to 2). The total NIHSS score is calculated by summing individual component scores. The max total score on NIHSS is 42 and the level of stroke severity as measured by the overall NIHSS score ranges from 0 (normal, no stroke) to 42 (severe stroke).
  The mean percent change from baseline is being reported; the greater the negative value, the better the outcome.
Time Frame: Baseline up to Day 84 post non-hemorrhagic ischemic stroke
Population: National Institutes of Health Stroke Scale (NIHSS) Score was assessed in the Primary Analysis population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | All Participants
Number analyzed (Participants) | 113
percent change
  Day 3 | -16.8 (30.94)
  Day 7 | -30.3 (40.33)
  Day 28: number analyzed (Participants) | 10
  Day 28 | -52.6 (57.21)
  Day 56: number analyzed (Participants) | 96
  Day 56 | -63.0 (43.60)
  Day 84: number analyzed (Participants) | 97
  Day 84 | -73.3 (30.66)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from baseline up to Day 84 post non-hemorrhagic ischemic stroke.
Description: This was an observational study and no study drug was administered; therefore, safety events were not assessed in this study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/120
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No